CLINICAL TRIAL: NCT02945657
Title: Protocol MEDI-MM36-206: A Phase 2 Multi-center, Open-label Study to Assess Pharmacokinetic Parameters and Safety of Topical MM36 (1%) in Pediatric Subjects 2 to < 18 Years of Age With Atopic Dermatitis Under Maximal Use Conditions
Brief Title: Pharmacokinetics and Safety of MM36 Topical Ointment in Pediatric Subjects With Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medimetriks Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MEDI-MM36-206
Record Dates: First submitted 2016-10-21; First posted 2016-10-26 (Estimated); Results first posted 2018-11-19 (Actual); Last update posted 2018-11-19 (Actual); Status verified 2018-11

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — difamilast

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MM36 1% ointment (Experimental): MM36 topical ointment, 1%, applied twice daily for 28 days
  Interventions: Drug: MM36 topical ointment, 1%

INTERVENTIONS:
Drug: MM36 topical ointment, 1% — Twice daily application for 28 consecutive days
  Other Names: OPA-15406

SUMMARY:
The purpose of this study is to assess the pharmacokinetic parameters and safety of topical MM36 (OPA-15406) ointment in pediatric subjects with atopic dermatitis under maximal use conditions.

DETAILED DESCRIPTION:
This is a multi-center, open-label study to assess the degree of systemic exposure and safety of MM36 1% ointment following 4 weeks of twice daily dosing under maximal-use conditions in pediatric subjects with atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 2 to <18 years of age
* Diagnosis of atopic dermatitis (AD)
* AD affecting ≥ 35% body surface area (BSA) if 2 to < 12 years of age or ≥ 25% if subject is ≥ 12 years of age (excluding scalp and venous access areas)

Exclusion Criteria:

* Active or acute viral skin infection
* History of recurrent bacterial infection
* Malignancy
* Clinically significant history or physical findings that may pose a health risk to subject or may have an impact on study assessments

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2016-10; Primary Completion 2017-06-08 (Actual); Study Completion 2017-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Noah Rosenberg, MD, Study Director — Medimetriks Pharmaceuticals, Inc
Locations (12):
- United States (10):
  - Medimetriks Investigational Site, Fremont, California
  - Medimetriks Investigational Site, Irvine, California
  - Medimetriks Investigational Site, San Diego, California
  - Medimetriks Investigational Site, Miami, Florida
  - Medimetriks Investigational Site, Saint Joseph, Missouri
  - Medimetriks Investigational Site, Portland, Oregon
  - Medimetriks Investigational Site, Austin, Texas
  - Medimetriks Investigational Site, Houston, Texas
  - Medimetriks Investigational Site, Norfolk, Virginia
  - Medimetriks Investigational Site, Spokane, Washington
- Medimetriks Investigational Site, San Pedro Sula, Honduras
- Medimetriks Investigational Site, Panama City, Panama

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- MM36 Topical Ointment, 1%: MM36 topical ointment, 1%, applied twice daily for 28 days
Period: Overall Study
Arm/Group | MM36 Topical Ointment, 1%
Started | 32
Completed | 28
Not Completed | 4
Not completed — Adverse Event | 1
Not completed — Withdrawal by Parent/Guardian | 3

BASELINE CHARACTERISTICS:
Arm/Group | MM36 Topical Ointment, 1%
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 32
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.9 (4.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 17
  More than one race | 7
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15
  Panama | 11
  Honduras | 6
Percentage of Body Surface Area (BSA) Involved [Mean (Standard Deviation); unit: %] | 43.7 (13.25)

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of MM36
Description: Maximum observed plasma concentration of MM36 on Day 1
Time Frame: Pre-dose (0 hour), 1, 4, and 8 hours post-dose on Day 1
Population: Pharmacokinetic (PK) population included participants in the Safety Population with PK Data
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- MM36 Topical Ointment, 1%: MM36 topical ointment, 1%, applied twice daily for 15 days
Arm/Group | MM36 Topical Ointment, 1%
Number analyzed (Participants) | 31
ng/mL | 23.1 (23.4)

2. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of MM36
Description: Maximum observed plasma concentration of MM36 after two weeks of twice daily application (steady state)
Time Frame: Pre-dose (0 hour), 1, 4, and 8 hours post-dose on Day 15
Population: Pharmacokinetic (PK) population included participants in the Safety Population with PK Data
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | MM36 Topical Ointment, 1%
Number analyzed (Participants) | 31
ng/mL | 16.9 (21.9)

3. Primary Outcome: Time of Maximum Observed Plasma Concentration (Tmax) of MM36
Description: Time of Maximum Observed Plasma Concentration (Tmax) of MM36 on Day 1
Time Frame: Pre-dose (0 hour), 1, 4, and 8 hours post-dose on Day 1
Population: Pharmacokinetic (PK) population included participants in the Safety Population with PK Data
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | MM36 Topical Ointment, 1%
Number analyzed (Participants) | 31
hours | 4.22 (2.02)

4. Primary Outcome: Time of Maximum Observed Plasma Concentration (Tmax) of MM36
Description: Time of Maximum Observed Plasma Concentration (Tmax) of MM36 on Day 15
Time Frame: Pre-dose (0 hour), 1, 4, and 8 hours post-dose on Day 15
Population: Pharmacokinetic (PK) population included participants in the Safety Population with PK Data
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | MM36 Topical Ointment, 1%
Number analyzed (Participants) | 31
hours | 3.80 (2.24)

5. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero To the Time of Last Quantifiable Plasma Concentration of MM36
Description: Area Under the Plasma Concentration-time Curve from Time Zero To the time of Last Quantifiable Plasma Concentration of MM36 on Day 1
Time Frame: Pre-dose (0 hour), 1, 4, and 8 hours post-dose on Day 1
Population: Pharmacokinetic (PK) population included participants in the Safety Population with PK Data
Measure: Mean (Standard Deviation); unit: ng·hr/mL
Arm/Group | MM36 Topical Ointment, 1%
Number analyzed (Participants) | 31
ng·hr/mL | 107 (94.1)

6. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero To the Time of Last Quantifiable Plasma Concentration of MM36
Description: Area Under the Plasma Concentration-Time Curve From Time Zero To the time of Last Quantifiable Plasma Concentration of MM36 on Day 15
Time Frame: Pre-dose (0 hour), 1, 4, and 8 hours post-dose on Day 15
Population: Pharmacokinetic (PK) population included participants in the Safety Population with PK Data
Measure: Mean (Standard Deviation); unit: ng·hr/mL
Arm/Group | MM36 Topical Ointment, 1%
Number analyzed (Participants) | 31
ng·hr/mL | 86.2 (79.6)

7. Secondary Outcome: Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Time Frame: up to 4 weeks
Population: Safety population included all subjects in the Intent to treat (ITT) population who had at least one post-baseline safety assessment
Measure: Number; unit: participants
Arm/Group | MM36 Topical Ointment, 1%
Number analyzed (Participants) | 31
participants
  No AE | 24
  AE | 7
  SAE | 0

8. Secondary Outcome: Treatment-Emergent Adverse Events (AEs) According to Severity
Description: Number of Participants With Treatment-Emergent Adverse Events (AEs) According to Severity. Adverse events were classified according to severity as: mild - an event that is usually transient in nature and generally not interfering with normal activities; moderate - an event that is sufficiently discomforting to interfere with normal activities; severe - an event that is incapacitating with inability to work or do usual activity or inability to work or perform normal daily activity.
Time Frame: up to 4 weeks
Population: Safety population included all subjects in the ITT population who had at least one post-baseline safety assessment
Measure: Number; unit: participants
Arm/Group | MM36 Topical Ointment, 1%
Number analyzed (Participants) | 31
participants
  None | 24
  Mild | 6
  Moderate | 1
  Severe | 0

9. Secondary Outcome: Application Site Adverse Events (AEs)
Description: Number of Participants With Application Site Adverse Events (AEs)
Time Frame: up to 4 weeks
Population: Safety population included all subjects in the ITT population who had at least one post-baseline safety assessment
Measure: Number; unit: participants
Arm/Group | MM36 Topical Ointment, 1%
Number analyzed (Participants) | 31
participants
  None | 29
  Application site pain | 1
  Application site rash | 1

10. Secondary Outcome: Application Site Adverse Events (AEs) According to Severity
Description: Number of Participants With Application Site Adverse Events (AEs) According to Severity. Adverse events were classified according to severity as: mild - an event that is usually transient in nature and generally not interfering with normal activities; moderate - an event that is sufficiently discomforting to interfere with normal activities; severe - an event that is incapacitating with inability to work or do usual activity or inability to work or perform normal daily activity.
Time Frame: up to 4 weeks
Population: Safety population included all subjects in the ITT population who had at least one post-baseline safety assessment
Measure: Number; unit: participants
Arm/Group | MM36 Topical Ointment, 1%
Number analyzed (Participants) | 31
participants
  None | 29
  Mild | 1
  Moderate | 1
  Severe | 0

11. Secondary Outcome: Clinically Meaningful Laboratory Test Median Changes From Baseline
Description: Number of Participants With Clinically Meaningful Laboratory Test Median Changes From Baseline. Clinical meaningfulness of laboratory test changes was determined at the investigator's discretion.
Time Frame: Day 29
Population: Safety population included all subjects in the ITT population who had at least one post-baseline safety assessment
Measure: Number; unit: participants
Arm/Group | MM36 Topical Ointment, 1%
Number analyzed (Participants) | 31
participants | 0

12. Secondary Outcome: Clinically Meaningful Vital Sign Median Changes From Baseline
Description: Number of Participants With Clinically Meaningful Vital Sign Median Changes From Baseline. Clinical meaningfulness of vital sign changes was determined at the investigator's discretion.
Time Frame: Day 29
Population: Safety population included all subjects in the ITT population who had at least one post-baseline safety assessment
Measure: Number; unit: participants
Arm/Group | MM36 Topical Ointment, 1%
Number analyzed (Participants) | 31
participants | 0

13. Secondary Outcome: Clinically Meaningful ECG Median Changes From Baseline to Day 15
Description: Number of Participants With Clinically Meaningful ECG Median Changes from Baseline. Clinical meaningfulness of ECG changes was determined at the investigator's discretion.
Time Frame: Day 15
Population: Safety population included all subjects in the ITT population who had at least one post-baseline safety assessment
Measure: Number; unit: participants
Arm/Group | MM36 Topical Ointment, 1%
Number analyzed (Participants) | 31
participants | 0

14. Secondary Outcome: Clinically Meaningful ECG Median Changes From Baseline to Day 29
Description: as for outcome 13
Time Frame: Day 29
Population: Safety population included all subjects in the ITT population who had at least one post-baseline safety assessment
Measure: Number; unit: participants
Arm/Group | MM36 Topical Ointment, 1%
Number analyzed (Participants) | 31
participants | 0

ADVERSE EVENTS:
Time Frame: up to 4 weeks
Arm/Group | MM36 Topical Ointment, 1%
All-Cause Mortality (participants affected / at risk) | 0/31
Serious Adverse Events (participants affected / at risk) | 0/31
Other Adverse Events (participants affected / at risk) | 7/31
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MM36 Topical Ointment, 1% (N=31)
Vomiting (Gastrointestinal disorders) | 1 (1)
Application site pain (General disorders) | 1 (1)
Application site rash (General disorders) | 1 (1)
Influenza like illness (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Eosinophil count increased (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Since the study is part of a multi-center study and an independent publication that will incorporate multi-center trial data is anticipated, Institution agrees not to independently publish its results of the study if such publication is published within 12 months from completion of the study. The Institution and Investigator agree not to publish the results of the study without prior written consent of the Sponsor, which consent may be withheld by Sponsor for any or no reason.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-05-18): https://cdn.clinicaltrials.gov/large-docs/57/NCT02945657/SAP_000.pdf
  • Study Protocol (2017-01-30): https://cdn.clinicaltrials.gov/large-docs/57/NCT02945657/Prot_001.pdf